CLINICAL TRIAL: NCT01827306
Title: Effectiveness of Biofreeze® on Shoulder Pain and In-office Exercise Performance: A Preliminary Pilot Study
Brief Title: Effectiveness of Biofreeze® on Shoulder Pain and In-office Exercise Performance
Acronym: BFShld01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sport and Spine Rehab Clinical Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SSR01
Record Dates: First submitted 2013-04-02; First posted 2013-04-09 (Estimated); Results first posted 2016-02-09 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-01

CONDITIONS: Shoulder Pain
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Biofreeze (Active Comparator): Apply 5 minutes before therapy by applying a small coin sized amount to the painful area. Subjects will then complete a standard shoulder therapy program.
  Interventions: Drug: Biofreeze
- Control (No Intervention): Subjects in this arm will complete a standard shoulder therapy program as normal, with no intervention.

INTERVENTIONS:
Drug: Biofreeze
  Arms: Biofreeze

SUMMARY:
Biofreeze® is a topical analgesic, frequently used in the office or given to a patient for home use as a way to mitigate pain during the course of treatment. Rehabilitative exercises are considered an important component of care for shoulder pain patients, although pain can be a limiting factor in the advancement of rehabilitation. The purpose of this study is to evaluate the addition of Biofreeze® to an in-office group of shoulder pain patients to determine its impact on pain reduction. Methods: Patients 18-64 years old with mechanical shoulder pain who are candidates for standard shoulder therapy will be randomized into two groups (N=20). The Control group (N=10) will receive standard shoulder therapy alone while the Intervention group (N=10) will receive standard shoulder therapy plus Biofreeze® just prior to initiating the in-office exercise program. Values of pain (NPRS) and disability (ASES) will be recorded at baseline, 2 weeks, and 4 weeks. Hypotheses will be addressed by repeated measures ANOVAs within and between group, time, and interaction main effects. Clinical Relevance: Progression of therapeutic exercises can be limited by pain and the associated disability. The ability to decrease shoulder pain and disability with a topical analgesic will allow health care professionals to advance patients through a therapeutic exercise program without the restriction of pain. In turn, patients will correct the underlying condition of their shoulder pain at a faster rate.

ELIGIBILITY:
Inclusion Criteria:

* 18-64 years old
* mechanical shoulder pain
* candidates for conservative care

Exclusion Criteria:

* pregnancy
* radicular symptoms
* not a candidate for conservative care
* history of recent shoulder surgery

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2013-03; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jay Greenstein, DC, Principal Investigator — Sport and Spine Rehab Clinical Research Foundation
Locations (1):
- Sport & Spine Rehab, Rockville, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Biofreeze: Apply 5 minutes before therapy by applying a small coin sized amount to the painful area. Subjects will then complete a standard shoulder therapy program.
  Biofreeze
- Control: Subjects in this arm will complete a shoulder therapy program as normal, with no intervention.
Period: Overall Study
Arm/Group | Biofreeze | Control
Started | 21 | 13
Completed | 10 | 8
Not Completed | 11 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Biofreeze | Control | Total
Number analyzed (Participants) | 21 | 13 | 34
Age, Continuous [Mean (Full Range); unit: years] | 42.19 [26 to 65] | 35.23 [19 to 49] | 39.53 [19 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 6 | 20
  Male | 7 | 7 | 14
Region of Enrollment [Number; unit: participants]
  United States | 21 | 13 | 34

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline of American Shoulder and Elbow Surgeons (ASES) Questionnaire at 2 Weeks
Description: The American Shoulder and Elbow Surgeons (ASES) Questionnaire is a self-report questionnaire measuring pain and disability. It is measured from 0 to 100, 0 being completely disabled and 100 being pain free and normal function. The total score is calculated using the following equation: (10-NPRS) x 5 = __ + (5/3) x Cumulative ADL Score
Time Frame: 2 weeks
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Biofreeze | Control
Number analyzed (Participants) | 10 | 8
units on a scale | 72.6 [55 to 83] | 68.75 [27 to 95]

2. Primary Outcome: Change From Baseline of Numeric Pain Rating Scale (NPRS) at 2 Weeks
Description: The Numeric Pain Rating Scale (NPRS) is a self-report scale measuring pain. It is measured from 0 to 10, 0 being pain free and 10 being the worse imaginable pain.
Time Frame: 2 weeks
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Biofreeze | Control
Number analyzed (Participants) | 10 | 8
units on a scale | 2.9 [2 to 5] | 3.75 [0 to 8]

3. Primary Outcome: Change From Baseline of American Shoulder and Elbow Surgeons (ASES) Questionnaire at 4 Weeks
Description: as for outcome 1
Time Frame: 4 weeks
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Biofreeze | Control
Number analyzed (Participants) | 10 | 8
units on a scale | 74.4 [47 to 100] | 77.13 [25 to 98]

4. Primary Outcome: Change From Baseline of Numeric Pain Rating Scale (NPRS)at 4 Weeks
Description: as for outcome 2
Time Frame: 4 weeks
Measure: Mean (Full Range); unit: units on a scale, from 0 to 10
Arm/Group | Biofreeze | Control
Number analyzed (Participants) | 10 | 8
units on a scale, from 0 to 10 | 2.6 [0 to 6] | 2.63 [0 to 8]

ADVERSE EVENTS:
Arm/Group | Biofreeze | Control
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/13
Other Adverse Events (participants affected / at risk) | 0/21 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No